CLINICAL TRIAL: NCT01390376
Title: DAAOI-1 Treatment for Treatment-resistant Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Collaborators: Department of Health, Executive Yuan, R.O.C. (Taiwan) (Other Government)
Responsible Party: Principal Investigator, Hsien-Yuan Lane, Departement of psychiatry, China Medical University Hospital, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DOH99-TD-I-111-TM001
Record Dates: First submitted 2011-07-07; First posted 2011-07-11 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; NMDA; DAAOI; Clozapine resistant schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- BE 1 (Experimental): DAAOI-1 1g
  Interventions: Drug: DAAOI-1
- BE 2 (Experimental): DAAOI-1 2g
  Interventions: Drug: DAAOI-1
- starch pill (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: DAAOI-1 — DAAOI-1 1g
  Arms: BE 1
Drug: DAAOI-1 — DAAOI-1 2g
  Arms: BE 2
Drug: placebo — starch pill
  Arms: starch pill

SUMMARY:
Pharmacotherapy for schizophrenia has limitations such as residual positive and negative symptoms, cognitive deficits and intolerable side effects. Refractory schizophrenia (particularly clozapine-resistant) is still a difficult clinical issue at present. According to the N-methyl-D-aspartate (NMDA) hypothesis, adjuvant NMDA-enhancing agents may have therapeutic benefit. DAAOI-1, a D-amino acid oxidase (DAAO) inhibitor, is a NMDA-enhancing agents.

The aim of this project is to examine the effectiveness and safety of DAAOI-1 adjuvant treatment for clozapine-resistant refractory schizophrenia patients in a randomized, double-blind, placebo - controlled trial.

DETAILED DESCRIPTION:
Pharmacotherapy for schizophrenia has limitations such as residual positive and negative symptoms, cognitive deficits and intolerable side effects. Refractory schizophrenia (particularly clozapine-resistant) is still a difficult clinical issue at present. Among schizophrenia patients, around 20-25%are treatment-resistant. According to the N-methyl-D-aspartate (NMDA) hypothesis, many clinical trials on NMDA-enhancing agents were studied. Adjuvant NMDA-enhancing agents, including glycine, D-amino acids (D-serine, D-alanine), and sarcosine (a glycine transporter I inhibitor), revealed beneficial but limited efficacy for positive and negative symptoms. The investigators recently started to study the potential of DAAOI-1, a D-amino acid oxidase (DAAO) inhibitor which can elevate synaptic concentration of D-amino acids.

The aims of this project is to examine the effectiveness and safety of DAAOI-1 adjuvant treatment for clozapine-resistant refractory schizophrenia patients in a randomized, double-blind, placebo - controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Fulfilled the DSM-IV criteria of schizophrenia
* Poor responder of clozapine: a 12-week treatment without satisfactory response: a minimal total score of 70 on the Positive and Negative Syndrome Scale (PANSS) (Kay 1987), and a minimal total score of 40 on the Scale for the Assessment of Negative Symptoms (SANS) (Andreasen 1983).
* Agree to participate in the study and provide informed consent

Exclusion Criteria:

* Meet DSM-IV criteria of other AXIS I disorder, current substance dependence or mental retardation
* Serious medical or neurological illness
* Pregnancy or lactation
* Use of depot antipsychotic in the past 6 months
* Inability to follow protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
The severity of psychiatric symptoms | week 0, 2, 4, 6
  The severity of psychiatric symptoms will be assessed by:
  1. Positive and Negative Syndrome Scale(PANSS)
  2. Assessment of Negative symptoms(SANS)
  3. Global assessment of function(GAF)
  4. Quality of life scale(QOL)

SECONDARY OUTCOMES:
PANSS subscales | week 0,2,4,6
  score changes
Hamilton Depression Rating Scale (HAMD) | Week 0,2,4, 6
Cognitive function | week 0, 6
  7 domains of Measurement and Treatment Research to Improve Cognition in Schizophrenia" [MATRICS]

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry, China Medical University Hospital, Taichung, Taiwan